CLINICAL TRIAL: NCT06145412
Title: A Phase II Trial of Xevinapant in Combination With Post-Operative Cisplatin and Radiotherapy for High Risk Head and Neck Cancer
Brief Title: A Study of Xevinapant With Cisplatin and Radiation Therapy After Surgery in People With Head and Neck Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-044
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Head and Neck Cancer
Keywords: Xevinapant; Cisplatin; Radiotherapy; 23-044
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Cisplatin

STUDY DESIGN:
Intervention Model Description: This is a single arm phase II.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Xevinapant in Combination with Post-Operative Cisplatin and Radiotherapy (Experimental): The study will consist of three phases: 2) concurrent radiation, cisplatin, and xevinapant, and 3) adjuvant xevinapant. Concurrent Chemoradiation Subjects will undergo FDG PET/CT simulation and standard radiation treatment planning. FDG PET/CT (Simulation or diagnostic) will also be utilized to rule out distant metastases. Subjects who meet criteria for the treatment phase will undergo standard of care adjuvant radiation (60-70 Gy administered in 2 Gy fractions) with concurrent cisplatin (2-3 cycles, with 100mg/m2 per cycle q3 weeks), and xevinapant (oral dose of 200mg per day on days 1-14 every 21 days for 3 cycles) Adjuvant Phase After completion of concurrent chemoradiation, patients will undergo an additional 3 cycles of xevinapant (oral dose of 200mg per day on days 1-14 every 21 days for 3- cycles)
  Interventions: Drug: Xevinapan; Drug: Cisplatin; Radiation: External beam

INTERVENTIONS:
Drug: Xevinapan — Xevinapant (oral dose of 200mg per day on days 1-14 every 21 days for 3 cycles)
Drug: Cisplatin — Cisplatin (2-3 cycles, with 100mg/m2 per cycle q3 weeks)
Radiation: External beam — 60 - 66 Gy in 2 Gy fractions for patients without gross disease and 70 Gy for patients with early recurrence) with concurrent cisplatin (40 mg/m2 once weekly)

SUMMARY:
The purpose of this study is to test whether treatment with Xevinapant added to standard chemoradiation after surgery is an effective treatment for people with high-risk head and neck cancers.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 on the day of signing of the consent form
* ECOG 0-1
* Able to swallow liquids or has an adequately functioning feeding tube, gastrostomy, or jejunostomy placed
* Squamous cell carcinoma of the head and neck (excluding lip) *

  o Eligible primary tumor sites will include the maxillary sinus, oral cavity, HPV-negative oropharynx, larynx, and hypopharynx.
* Gross total resection of known disease at the time of surgery within 10 weeks of registration. All efforts will be made to begin treatment within 6 weeks of surgery.
* At least one of the following criteria

  * Close surgical margin (<5mm) AND ≥2 additional intermediate risk factors (T3 or T4, multiple lymph nodes, LVI, PNI)
  * Positive margins not eligible for re-resection (defined as <1mm)
  * Extranodal extension
  * Evidence of early gross recurrence on radiation planning scans after definitive intent surgical resection Patients with evidence of gross locoregional disease at the time of radiation are strongly advised to have biopsy confirmation. This requirement may be waived by the PI or the co-PIs. If a biopsy is not performed, patients must meet one of the other entry criteria (close surgical margin and 2 or more additional intermediate risk factors; positive margins not eligible for re-resection; extranodal extension).
* Adequate hematologic, renal, and hepatic function as indicated by:

  * Absolute neutrophil count ≥ 1 500 cells/μL
  * Platelets ≥ 100 000 cells/μL
  * Hemoglobin ≥ 9.0 g/dL (blood transfusions during screening are permitted)
  * AST and ALT ≤ 3.0 × upper limit of normal (ULN)
  * Total bilirubin ≤ 1.5 × ULN (up to 2.0 × ULN is allowed if the direct bilirubin level is normal, and the elevation is limited to indirect bilirubin).
* Adequate renal function within 30 days prior to registration, defined as follows:

Creatinine clearance (CC) ≥ 60 ml/min determined by 24-hour collection or estimated by Cockcroft-Gault formula:

* CCr male = [(140 - age) x (wt in kg)] [(Serum Cr mg/dl) x (72)]
* CCr female = 0.85 x (CrCl male) Women of childbearing potential (according to recommendations of the Clinical Trial Facilitation Group) must have a negative serum pregnancy test at screening and must not be breastfeeding.

  * Women of childbearing potential must agree to use highly effective contraceptive method(s). from ICF signature to 6 months after the last administration of chemotherapy or 3 months after last dose of xevinapant, whichever is the latest.
  * Non-sterilized males who are sexually active with a female partner of childbearing potential must agree to use condom and spermicide from ICF signature to 6 months after the last administration of chemotherapy or 3 months after the last dose of xevinapant, whichever is the latest.
  * Because male condom and spermicide is not a highly effective contraception method, it is required that female partners of a male study subject use highly effective contraceptive method(s) throughout this period.
  * Male subjects must refrain from donating sperm during the clinical study and for 6 months after the last administration of chemotherapy or 3 months after the last dose of xevinapant, whichever is the latest.
  * If not done previously, cryopreservation of sperm prior to receiving chemotherapy or xevinapant is advised to male patients with a desire to have children.

Exclusion Criteria:

* Metastatic disease

  * Prior head and neck radiation
  * Peripheral Neuropathy ≥ grade 2
  * Hearing Impairment ≥ grade 2
  * On-going wound infection, fistula, flap failure
  * Use within 14 days prior to randomization or requirement for ongoing treatment with any drug(s) on the prohibited medication list (see below).
  * Known history of infection with HIV. If unknown history of HIV, an HIV screening test is to be performed and subjects with positive serology for HIV-1/2 must be excluded.
  * Known chronically active HBV or HCV infection. If unknown status, the following tests are to be performed and subjects with positive serology must be excluded:

    * HBV screening tests: both HBV sAg and Anti-HepB core IgG.
    * HCV screening tests: both HCV-antibody and positive viral load HCV-RNA by PCR.
    * Other infections (viral and/or bacterial and/or mycotic) requiring systemic treatment.
  * Live-attenuated vaccinations within 30 days prior to first investigational treatment administration.

Ongoing uncontrolled infection requiring intravenous antibiotic therapy within 1 week prior to randomization.

* Documented weight loss of >10% during the last 4 weeks prior to randomization (unless adequate measures are undertaken for nutritional support), OR plasmatic albumin <3.0 g/dL. No albumin transfusions are allowed within 2 weeks before randomization.
* Active uncontrolled inflammatory disease (including rheumatoid arthritis, systemic lupus erythematosus, Sjögren syndrome, severe extensive psoriasis, and other autoimmune diseases) requiring ongoing treatment with anti-TNF medication.
* Any concomitant medication known to prolong the QT interval that cannot be discontinued or replaced by safe alternative medication within 7 days prior to start of treatment.
* Known allergy to Xevinapant or any excipient known to be present in the formulation.
* Non-compensated or symptomatic liver cirrhosis (Child-Pugh score: B or C).
* Treatment with an investigational agent or use of an investigational device within 4 weeks of the first dose of study treatment.
* Known gastrointestinal disorder with clinically established malabsorption syndrome and major gastrointestinal surgery that may limit oral absorption.
* Active gastrointestinal bleeding, or any other uncontrolled bleeding requiring more than 2 red blood cell transfusions or 4 units of packed red blood cells within 4 weeks prior to randomization.
* Impaired cardiovascular function or clinically significant cardiovascular diseases, including any of the following:

  * Ongoing or history of uncontrolled or symptomatic ischemic myocardiopathy within 6 months prior to randomization.
  * Known left ventricular ejection fraction < 50%).
  * History of myocardial infarction, or severe/unstable angina, within 6 months prior to randomization.
  * New York Heart Association grade ≥ 3 congestive heart failure.
  * Congenital long QT syndrome.
  * Family history of long QT syndrome.
  * Symptomatic pulmonary embolism within 6 months prior to randomization.
  * Ongoing or known history of transient ischemic attacks or stroke within 6 months prior to randomization.
  * QTc using Fridericia's formula (QTcF) interval > 450 ms for males and > 470 ms for females Symptomatic pulmonary disease requiring continuous or intermittent oxygen supply.
* History of another malignancy within the last 3 years prior to randomization, with the exception of completely resected non-melanoma cell skin cancer outside the head and neck area or completely resected stage I breast cancer, or completely resected in-situ non-muscular invasive bladder, cervix and/or uterine carcinomas.
* Any ongoing condition or disorder, before randomization, including drug(s) or alcohol abuse, which in the judgment of the Investigator would make the patient inappropriate for entry into the study or precluding his/her ability to comply with study procedures.
* Lack of ability to understand and willingness to sign a written informed consent and complete questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-11-16 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 12 months
  Progression free survival will be defined as the time from the start of treatment to biopsyproven locoregional recurrence, distant tumor recurrence, or death. For patients without evidence of gross disease at registration, any locoregional progression will be considered a PFS event. For patients with gross disease at registration, progression-free survival will be determined based upon RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Overall survival | 3 years
  Overall survival will be defined as the time from treatment start to the time of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Yao Yu, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/